CLINICAL TRIAL: NCT00704249
Title: Randomized Multicenter Study to Compare Starting Nevirapine at the Full Dose With Dose Escalation in Patients Who Require Efavirenz to be Withdrawn Due to Adverse Reactions
Brief Title: VENICE Study Nevirapine Full Dose/Dose Escalation
Acronym: VENICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Trial Agency of HIV Study Group (Other)
Responsible Party: Esteban Ribera, Clinical Trial Agency of HIV Study Group
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GESIDA-4905
Record Dates: First submitted 2008-06-22; First posted 2008-06-24 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: HIV infection; nevirapine; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (2):
- 1 (Experimental): Full-dose nevirapine from baseline (200 mg bid).
  Interventions: Drug: nevirapine
- 2 (Active Comparator): Nevirapine with an increase in the initial dose (200 mg once daily for 14 days and 200 mg bid thereafter)
  Interventions: Drug: nevirapine

INTERVENTIONS:
Drug: nevirapine — Full-dose nevirapine from baseline (200 mg bid).
  Arms: 1
Drug: nevirapine — Nevirapine with an increase in the initial dose (200 mg once daily for 14 days and 200 mg bid thereafter)
  Arms: 2

SUMMARY:
This study aims to compare the trough plasma concentrations of nevirapine after 7 days of treatment at the full dose from baseline with dose escalation in patients taking efavirenz who switch to nevirapine due to neuropsychiatric adverse reactions.

DETAILED DESCRIPTION:
The prognosis for HIV infection changed radically after 1996 thanks to the arrival of protease inhibitors (PI), which, when combined with 2 nucleoside analogue reverse transcriptase inhibitors (NRTI) formed the so-called highly active antiretroviral therapy (HAART). HAART led to a considerable decrease in the incidence and mortality of opportunistic infections and made HIV infection a chronic condition and not necessarily the progressive, irreversible, and fatal disease it was before 1996. The initial euphoria led people to believe that HAART could cure the disease, but it was soon clear that eradication of the virus was impossible and that treatment would have to be continued indefinitely. Chronic treatment became more difficult because of the frequent onset of adverse events or extremely complex regimens with a high pill burden that had to be administered several times per day, often with dietary restrictions.1,2 In this context, adherence was difficult, efficacy was far from optimal, and the patient's quality of life was noticeably reduced. The subsequent appearance of non-nucleoside analogue reverse transcriptase inhibitors (NNRTI)-nevirapine and efavirenz-considerably improved some of the disadvantages of PIs. Today, the combination of 2 NRTIs and an NNRTI is considered the regimen of choice when starting antiretroviral therapy. Efavirenz is considered the gold standard for initial antiretroviral therapy and is widely used in clinical practice.

More than half of the patients who start treatment with efavirenz present adverse effects, although these are generally well tolerated and decrease with time. Approximately 3%-8% of patients have to suspend efavirenz due to adverse effects, which are mainly neuropsychiatric. In these cases, efavirenz is usually replaced by nevirapine.

Nevirapine is a substrate and potent inducer of the hepatic cytochrome P450 enzyme system (CYP3A4 and others) and continuous administration leads to progressive autoinduction of its own metabolism. The recommended dose is 200 mg every 12 hours. If this dose is administered from the start of treatment, the plasma concentrations reached during the first few days are much higher than those reached later. Therefore, and because the toxicity of nevirapine is associated with its plasma concentrations, the recommended initial dose is 200 mg/d for the first 14 days followed by 200 mg every 12 hours indefinitely. There are no specific recommendations on dosage when nevirapine replaces efavirenz; therefore, it is administered at increasing doses according to the summary of product characteristics.

Efavirenz is also a potent inducer of CYP3A4 and increases the metabolism of other drugs that use this metabolic pathway. Enzyme induction is by increased synthesis of the enzymes involved, with the result that, when the inducer is suspended, the enzyme induction effect persists for a few days until the excess enzymes are catabolized. Furthermore, the half-life of efavirenz is very long. Consequently, the plasma concentrations fall progressively for more than a week after the drug is withdrawn. Therefore, when efavirenz is replaced by nevirapine, the residual enzyme induction that persists might lead to a fall in the plasma concentrations of nevirapine. Given that NNRTIs have a low genetic barrier for the development of resistance, the fall in plasma concentrations of nevirapine for the 14 days during which it is administered at 200 mg/d can generate resistance mutations and virologic failure.

When efavirenz is switched for nevirapine, it is unknown whether nevirapine should be started at increasing standard doses (200 mg/d for the first 14 days plus 200 mg bid thereafter) or at the full dose (200 mg every 12 hours) as a consequence of the enzyme induction caused by efavirenz.

Currently available data do not enable us to make a recommendation on the dose with which treatment with nevirapine can be started in patients who required efavirenz to be withdrawn and for whom nevirapine was chosen as an alternative. Nevertheless, despite small sample sizes, preliminary studies suggest that this strategy could be effective and safe. Therefore, randomized clinical trials that enable us to evaluate this strategy appropriately are necessary

ELIGIBILITY:
Inclusion Criteria:

* Age ³ 18 years
* Chronic HIV-1 infection confirmed by Western blotting
* Patients treated with a HAART regimen containing efavirenz for a minimum of 15 days before the baseline visit
* Patients who present a neuropsychiatric adverse reaction to efavirenz (see list in Appendix D) and require it to be withdrawn.
* Ability of the patient to follow treatment during the period established
* Acceptance and signing of the informed consent document

Exclusion Criteria:

* Liver function test (AST, ALT, GGT) results > 3 times the upper limit of normal.
* Elevated creatinine levels (>1.5 mg/dL)
* CD4+ T-cell count > 400 cells/µL in men or > 250 cells/µL in women, unless the benefit outweighs the risk (warning in the summary of product characteristics) and always at the investigator's discretion
* HIV plasma viral load > 50 copies/mL in those patients who have been taking efavirenz for more than 3 months
* Suspected or confirmed resistance to efavirenz and/or nevirapine
* Patients who are currently taking a drug that might interfere in the absorption, distribution, or metabolism of nevirapine
* Presence of opportunistic infections and/or neoplasm during the 3 months before the start of participation in the trial
* Any medical condition(s) that, in the investigator's opinion, might interfere with the patient's ability to participate or fulfill the requirements of the present protocol
* Pregnancy
* Suspected primary infection of less than 6 months' duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a trough concentration of nevirapine in plasma within the therapeutic range (3000 to 8000 ng/mL) after 7 days of treatment. | 7 days

SECONDARY OUTCOMES:
The proportion of patients with a plasma viral load of less than 50 copies/mL will be obtained. The change in CD4+ T-cell count will also be measured from baseline to weeks 4 and 12. | 12 weeks
The proportion of patients who experience adverse events (proportion of patients with exanthema and proportion of patients with liver toxicity) | 4 weeks
Proportion of patients with resolution of the neuropsychiatric adverse reaction to efavirenz that led to it being withdrawn | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Ribera, Study Chair — Clinical Trial Agency of HIV Study Group
Locations (15):
- Spain (15):
  - Hospital General Alicante, Alicante, Alicante
  - Hospital General de Elche, Elche, Alicante
  - Hospital Germanas Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Santa Creu y Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Vall d´Hebrón, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Provincial Reina Sofía de Córdoba, Córdoba, Cordoba
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Virgen de la Victoria, Málaga, Malaga